CLINICAL TRIAL: NCT02753569
Title: Imaging NSCLC Treatment Response to Immunotherapy: Relating Inflammatory Activity on 18FDG PET to Tumour Specific Measures From DW-MRI
Brief Title: Imaging NSCLC Treatment Response to Immunotherapy
Status: Completed | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Nandita deSouza, Professor of Translational Imaging, Institute of Cancer Research, United Kingdom
Other Study IDs: CCR4364
Record Dates: First submitted 2016-04-20; First posted 2016-04-28 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Cancer
Keywords: Magnetic Resonance Imaging; PET/CT; non-small cell lung cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Imaging - DW-MRI
Radiation: FDG PET-CT

SUMMARY:
This feasibility study will aim to assess the potential for functional imaging biomarkers (18FDG PET-CT and DW-MRI) to differentiate immunotherapy induced inflammation, indicative of response from non-response in patients with stage IV non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
30 patients, recruited from within the PEAR Study (Phase 1 dose escalation of palliative radiotherapy with anti-PD1 antibody pembrolizumab in thoracic tumours) will be scanned both before and after receiving immunotherapy for NSCLC. Immunotherapy induced changes in tumour ADC on DW-MRI (a surrogate of apoptotic tumour cell death) will be compared with changes in near contemporaneous, anatomically co-registered 18FDG PET-CT SUV (a non-specific marker for GLUT expression and hence metabolic activity in both tumour and tumour infiltrating lymphocytes). For treatment response, an increase in ADC (reflecting apoptosis within the tumour) is expected, while 18FDG uptake is expected to decrease compared with baseline tumour uptake. In the presence of significant inflammatory cell recruitment, the investigators hypothesise a similar increase in ADC on DW-MRI but without associated reduction in 18FDG PET-CT SUV. Thus the relationship between the ADC change on DW-MRI and the 18FDG change should distinguish between response and non-response in the presence of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Recruited to PEAR: Phase 1 dose escalation of palliative radiotherapy with anti-PD1 antibody pembrolizumab in thoracic tumours Study

Exclusion Criteria:

* MRI incompatible metal implants
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with NSCLC requiring palliative radiotherapy to the chest and for which no curative therapy exists.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Changes in DW-MRI derived ADC | Duration of Study - 2 year
  Describing changes in DW-MRI derived ADC will provide data that may be used to differentiate immune mediated response from non-response in a future study of treatment responses following immunotherapy.
Changes in FDG PET/CT SUV | Duration of Study - 2 year
  Describing changes in 18FDG-PET SUV will provide data that may be used to differentiate immune mediated response from non-response in a future study of treatment responses following immunotherapy.

SECONDARY OUTCOMES:
Assess for differences in tumour volume using DW-MRI | Duration of Study - 2 year
  Assess for differences in tumor volume evaluated using DW-MRI. This will be used as a comparison against other modalities for assessing differences in tumour volume e.g. 18FDG PET-CT. CT is the current standard for radiotherapy target volumes in the chest and with the greater soft tissue delineation facilitated by MRI, comparison of the modalities is warranted.
Assess for differences in tumour volume using 18FDG PET-CT | Duration of Study - 2 year
  Assess for differences in tumor volume evaluated using 18FDG PET-CT. This will be used as a comparison against other modalities for assessing differences in tumour volume e.g. MRI. CT is the current standard for radiotherapy target volumes in the chest and with the greater soft tissue delineation facilitated by MRI, comparison of the modalities is warranted.
Assess correlation between DW-MRI derived ADC and FDG PET/CT SUV | Duration of Study - 2 year
  Assess the correlation between 18FDG PET Standardised Uptake Values and DW-MRI derived ADC values. Correlations between ADCmax and SUVmax; ADCmean and SUVmean; plus total lesion ADC and total lesion glycolysis will be explored. Recent reports of imaging biomarkers for defining radiotherapy 'dose painting' schedules have focussed on PET imaging and correlation of these parameters with DW-MRI is not yet established.
Ability to predict progression free time and overall survival using DW-MRI ADC | Duration of Study - 2 year
  Assess DW-MRI ADC, used alone or in combination with 18FDG SUV (before and after immunotherapy), for its ability to predict progression free and overall survivals following subsequent radiotherapy.
Ability to predict progression free time and overall survival using 18FDG SUV | Duration of Study - 2 year
  Assess 18FDG SUV, used alone or in combination with DW-MRI ADC (before and after immunotherapy), for their ability to predict progression free and overall survivals following subsequent radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom